CLINICAL TRIAL: NCT05926206
Title: A Multicenter Open-Label Dose Optimization Trial of Devimistat in Combination With Modified FOLFIRINOX in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Trial of Devimistat in Combination With Modified FOLFIRINOX in Patients With Metastatic Adenocarcinoma of the Pancreas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: based some additional data, we have decided to hold off this trial for now and will not be proceeding with this particular trial
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2022.126; HUM00228911 (Other: University of Michigan)
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — devimistat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- TiTE-CRM Dose Escalation (Experimental): Devimistat at Dose Level IV 2 hrs + modified FOLFIRINOX
  Interventions: Drug: Devimistat; Drug: Modified FOLFIRINOX
- Expansion Cohort A (Experimental): Devimistat 500 mg/m2 IV 2 hrs + modified FOLFIRINOX
  Interventions: Drug: Devimistat; Drug: Modified FOLFIRINOX
- Expansion Cohort B (Experimental): Devimistat at MTD IV 4 hrs + modified FOLFIRINOX
  Interventions: Drug: Devimistat; Drug: Modified FOLFIRINOX

INTERVENTIONS:
Drug: Devimistat — Escalation: Assigned dose level (mg/m2), IV over 120 minutes, Days 1 and 3 Cohort A: 500 mg/m2, IV over 120 minutes, Days 1 and 3 Cohort B: MTD mg/m2, IV over 240 minutes, Days 1 and 3
Drug: Modified FOLFIRINOX — Oxaliplatin- 85 mg/m2, IV over 120 minutes, day 1 Leucovorin/folinic acid- 400 mg/m2, IV over 90 minutes, day 1 Irinotecan- 150 mg/m2, IV over 90 minutes, day 1 5FU- 2400 mg/m2, IV over 42-48 hours after irinotecan, day 1

SUMMARY:
This protocol will enroll patients with metastatic pancreatic cancer to receive modified FOLFIRINOX plus devimistat. Patients will be enrolled with 1:1 randomization between Dose Escalation Cohort and Cohort A until required 20 patients have been enrolled on Cohort A following which randomization will end and patients will be enrolled without randomization to Dose Escalation Cohort and then subsequently to Cohort B.

ELIGIBILITY:
Eligibility Criteria:

* Histologically or cytologically confirmed metastatic stage IV adenocarcinoma of the pancreas
* No prior systemic treatment for advanced pancreatic adenocarcinoma. Prior adjuvant or neoadjuvant treatment is allowed provided it completed ≥ 6 months prior to disease recurrence. Palliative radiation therapy is allowed provided it completed ≥ 2 weeks prior to starting trial therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Age 18 years or greater
* Measurable disease determined using guidelines of Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must agree to use acceptable highly effective contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive(s), intrauterine hormone releasing system (IUS), bilateral tubal occlusion or vasectomized partner) starting at screening, during the study, and for 9 months after last study dose and must have a negative serum or urine pregnancy test during screening.
* Males with female partners (of childbearing potential) must agree to use double barrier contraceptive measure (a combination of male condom with either cap, diaphragm or sponge with spermicide) in addition to oral contraception, or avoidance of intercourse during the study and for 6 months after last study dose is received.
* At least 4 weeks from major surgery with resolution of any sequela to date of enrollment
* Laboratory values ≤2 weeks during screening must be: Platelet count ≥ 100,000 cells/mm3, Absolute neutrophil count ≥ 1500 cells/mm3, Hemoglobin > 9 g/dL, AST/ALT ≤ 3x upper limit of normal [ULN], or (≤ 5x ULN if liver metastasis present), Bilirubin ≤ 1.5x ULN, or (≤ 2.5 x ULN for subjects with Gilbert's syndrome), Albumin > 3 g/dL, Serum creatinine clearance CrCl > 30 mL/min per Cockcroft-Gault Formula, INR <1.5 unless on anticoagulants
* No evidence of active infection and no serious infection within the past 30 days. Patient must have completed antibiotic course.
* Mentally competent, ability to understand and willingness to sign the informed consent form and follow protocol requirements
* No known central nervous system metastasis or epidural tumor
* No known hypersensitivity to devimistat, platinum-based drugs, FOLFIRINOX treatment or any of their excipients
* Patients must not have received any other investigational systemic agent for any indication within the past 2 weeks prior to initiation of devimistat treatment
* No active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., Hemophilia A)
* Female patients must not be pregnant, have a positive pregnancy test, breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 9 months after the last dose of study treatment.
* Male patients must be willing to abstain from donating sperm during treatment and for 6 months after completion of study treatment
* No active heart disease including but not limited to myocardial infarction that is <3 months prior to registration, symptomatic congestive heart failure (NYHA class 3 or 4), symptomatic coronary artery disease, symptomatic angina pectoris
* No prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, in situ cancer, localized prostate cancer (Gleason score <8), or adequately treated cancer from which the patient has been disease-free for at least 3 years prior to registration.
* Patients must not be using strong CYP3A4 inducers or inhibitors (as listed in Appendix II: CYP3A4 Inducers or Inhibitors)
* No marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 470 milliseconds (ms) (CTCAE grade 1) using Fridericia's QT correction formula (i.e. QTcF); or history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).
* Patients must not have known reduced UGT1A1 or DPD activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicity during the first 15 days of devimistat in combination with modified FOLFIRINOX in the dose escalation cohort | 15 days post the start of combination therapy
  The maximum tolerated dose (MTD) will be determined based on dose limiting toxicity
Median Progression Free Survival (PFS) of devimistat plus modified FOLFIRINOX across all cohorts | up to 42 months after enrollment
  The PFS will be defined as time from date of initial treatment to date of radiological or clinical progression (leading to withdrawal from the study treatment), or death from any cause on study treatment, whichever comes first. Follow-up time will be censored at the date of last disease evaluation.

SECONDARY OUTCOMES:
Number of subjects with reported adverse events and reportable serious events | up to 25 months after enrollment
  To assess the safety and toxicity of the drug combination by reported adverse events and reportable serious events are defined by the study protocol (NCI Common Toxicity Criteria for Adverse Events (CTCAE) v5.0).
Overall Response Rate (ORR) of devimistat plus modified FOLFIRINOX | up to 42 months after enrollment
  ORR will be determined as per the RECISTv1.1 criteria
Overall Survival (OS) of devimistat plus modified FOLFIRINOX | up to 42 months after enrollment
  OS will be defined from the date of initial treatment to either date of death or censoring.
Overall Survival (OS) of devimistat plus modified FOLFIRINOX based on gender | up to 42 months after enrollment
  OS will be defined from the date of initial treatment to either date of death or censoring.
Duration of response (DoR) of devimistat plus modified FOLFIRINOX | up to 42 months after enrollment
  DoR will be measured from the start date of the best response achieved until the date of relapse (i.e., progression). Continuing responders will be right-censored as of the most recent date on which their response status had been assessed. DoR applies to only the patients who achieve either a complete response or a partial response.
To assess pharmacokinetics (Cmax) of devimistat | up to 42 months after enrollment
  The PK parameters of devimistat (and its metabolites, if appropriate), including but not limited to peak plasma concentration (Cmax) versus time curve from time 0 to t (AUC0-t)
To assess pharmacokinetics (AUCinf) of devimistat | up to 42 months after enrollment
  The PK parameters of devimistat (and its metabolites, if appropriate), including but not limited to area under the concentration versus time curve from time 0 to infinity (AUCinf)
To assess pharmacokinetics (t1/2) of devimistat | up to 42 months after enrollment
  The PK parameters of devimistat (and its metabolites, if appropriate), including but not limited to elimination half-life (t1/2)
To assess pharmacokinetics (tmax) of devimistat | up to 42 months after enrollment
  The PK parameters of devimistat (and its metabolites, if appropriate), including but not limited to time to reach the maximum plasma concentration (tmax)
To assess pharmacokinetics (CL) of devimistat | up to 42 months after enrollment
  The PK parameters of devimistat (and its metabolites, if appropriate), including but not limited to clearance (CL)
To assess pharmacokinetics (Vd) of devimistat | up to 42 months after enrollment
  The PK parameters of devimistat (and its metabolites, if appropriate), including but not limited to volume of distribution (Vd)
To determine the median Progression Free Survival (PFS) of devimistat plus modified FOLFIRINOX based on gender | up to 42 months after enrollment
  The PFS will be defined as time from date of initial treatment to date of radiological or clinical progression (leading to withdrawal from the study treatment), or death from any cause on study treatment, whichever comes first. Follow-up time will be censored at the date of last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators interested in data would email the study PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study publication
Access Criteria: Investigators interested in data would email the study PI